CLINICAL TRIAL: NCT06074588
Title: A Randomized, Open-label, Phase 3 Study of MK-2870 vs Chemotherapy (Docetaxel or Pemetrexed) in Previously Treated Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With EGFR Mutations or Other Genomic Alterations
Brief Title: Sacituzumab Tirumotecan (MK-2870) Versus Chemotherapy in Previously Treated Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With EGFR Mutations or Other Genomic Alterations (MK-2870-004)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-004; 2023-503539-16-00 (Registry Identifier: EU CT); jRCT2031240108 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1287-4913 (Registry Identifier: UTN)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Anaplastic lymphoma kinase (ALK); Antibody-drug conjugate (ADC); Epidermal growth factor receptor (EGFR); Trophoblast cell-surface antigen 2 (TROP2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab tirumotecan (Experimental): Participants will receive 4 mg/kg of sacituzumab tirumotecan via intravenous (IV) infusion on Days 1, 15 and 29 of each 6-week cycle. Additionally, participants receive diphenhydramine (or equivalent), an H2 antagonist of investigator's choice, acetaminophen (or equivalent), and dexamethasone (or equivalent) per each drug's product label prior to the first 4 infusions of sacituzumab tirumotecan. At subsequent infusions, the H2 antagonist and dexamethasone are optional, at the discretion of the investigator.
  Interventions: Biological: Sacituzumab tirumotecan
- Chemotherapy (Active Comparator): Participants will receive 75 mg/m^2 of docetaxel or 500 mg/m^2 of pemetrexed by IV infusion on Days 1 and 22 of every 6-week cycle.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — 4 mg/kg of MK-sacituzumab tirumotecan by IV infusion
  Other Names: SKB264, MK-2870
  Arms: Sacituzumab tirumotecan
Drug: Docetaxel — 75 mg/m^2 of docetaxel by IV Infusion
  Other Names: TAXOTERE®
  Arms: Chemotherapy
Drug: Pemetrexed — 500 mg/m^2 of pemetrexed by IV infusion
  Other Names: ALIMTA®
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to evaluate sacituzumab tirumotecan versus chemotherapy (docetaxel or pemetrexed) for the treatment of previously-treated non-small cell lung cancer (NSCLC) with exon 19del or exon 21 L858R EGFR mutations (hereafter referred to as EGFR mutations or EGFR-mutated) or any of the follow genomic alterations: ALK gene rearrangements, ROS1 rearrangements, BRAF V600E mutations, NTRK gene fusions, MET exon 14 skipping mutations, RET rearrangements, or less common EGFR point mutations of exon 20 S768I, exon 21 L861Q, or exon 18 G719X mutations. The primary hypotheses are that sacituzumab tirumotecan is: (1) superior to chemotherapy with respect to progression-free survival (PFS) per RECIST 1.1 as assessed by BICR in NSCLC with EGFR mutations; and (2) superior to chemotherapy with respect to overall survival (OS) in NSCLC with EGFR mutations.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Histologically- or cytologically-documented advanced (Stage III not eligible for resection or curative radiation) or metastatic non-squamous NSCLC with specific mutations.
* Documentation of locally assessed radiological disease progression while on or after last treatment based on Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1.
* Participants with genome mutations must have received 1 or 2 prior lines of epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI), including a third generation TKI for participants with a T790M mutation; and 1 platinum-based therapy after progression on or after EGFR TKI.
* Measurable disease per RECIST 1.1 as assessed by the local site investigator.
* Archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated has been provided
* Participants who have AEs due to previous anticancer therapies must have recovered to Grade ≤1 or baseline.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy.
* Have an ECOG performance status of 0 or 1 within 3 days before randomization.

Exclusion Criteria:

* Has predominantly squamous cell histology NSCLC.
* Has mixed tumor(s) with small cell elements.
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease.
* Has Grade ≥2 peripheral neuropathy.
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or corneal disease that prevents/delays corneal healing.
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease.
* Has an EGFR T790M mutation and has not received a third generation EGFR TKI (eg, osimertinib).
* Received prior systemic anticancer therapy including investigational agents within 4 weeks or 5 half-lives (whichever is shorter) before randomization.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Completed palliative radiotherapy within 7 days of the first dose. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.
* Received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study intervention.
* Received prior treatment with a trophoblast cell-surface antigen 2 (TROP2)-targeted antibody-drug conjugate (ADC).
* Received prior treatment with a topoisomerase I-containing ADC.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Active infection requiring systemic therapy.
* History of noninfectious pneumonitis/ILD that required steroids or has current pneumonitis/ILD.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are clinically stable, radiologically stable for at least 4 weeks and do not require glucocorticoids for at least 14 days prior to randomization.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2030-03-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) of Participants with NSCLC with Epidermal Growth Factor Receptor (EGFR) Mutations | Up to approximately 35 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review (BICR) or death due to any cause, whichever occurs first.
Overall Survival (OS) of Participants with NSCLC with EGFR mutations | Up to approximately 41 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
PFS of All Participants with NSCLC | Up to approximately 35 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.
OS of All Participants with NSCLC | Up to approximately 41 months
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) of Participants with NSCLC with EGFR Mutations | Up to approximately 35 months
  ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. based on BICR in NSCLC with EGFR mutations.
ORR of All Participants with NSCLC | Up to approximately 35 months
  ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. based on BICR in all participants with NSCLC.
Duration of Response (DOR) of All Participants with NSCLC | Up to approximately 6 years
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR in all participants with NSCLC, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Change in Score from Baseline in Global Health Status/QoL Score (European Organisation for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-Core 30 [QLQ-C30] Items 29 and 30) | Baseline and up to approximately 48 weeks
  The EORTC QLQ-C30 is a questionnaire to assess the overall health status and quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status and quality of life. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change in Score from Baseline in Dyspnea Score (EORTC QLQ-C30 Item 8) | Baseline and up to approximately 48 weeks
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea. The change from baseline in the dyspnea (EORTC QLQ-C30 Item 8) score will be presented.
Change in Score from Baseline in Cough (EORTC Quality of Life Questionnaire-Lung Cancer 13 [QLQ-LC13] Item 31) | Baseline and up to approximately 48 weeks
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in cough (EORTC QLQ-LC13 Item 31) score will be presented. A lower score indicates a better outcome.
Change in Score from Baseline in Chest Pain (EORTC QLQ-LC13 Item 40) | Baseline and up to approximately 48 weeks
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented. A lower score indicates a better outcome.
Time to Deterioration (TTD) from Baseline in Global Health Status/QoL Score (EORTC QLQ-C30 Items 29 and 30) | Up to approximately 48 weeks
  The EORTC QLQ-C30 is a questionnaire to assess the overall health status and quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status and quality of life. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Items 29 and 30 will be presented.
TTD from Baseline in Dyspnea Score (EORTC QLQ-C30 Item 8) | Up to approximately 48 weeks
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicates a worse level of dyspnea. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-C30 Item 8 will be presented.
TTD from Baseline in Cough (EORTC Quality of Life Questionnaire-Lung Cancer 13 [QLQ-LC13] Item 31) | Up to approximately 48 weeks
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate more frequent coughing and a worse outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-LC13 Item 31 will be presented.
Time to Deterioration from Baseline in Chest Pain (EORTC QLQ-LC13 Item 40) | Up to approximately 48 weeks
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate worse level of chest pain. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline. TTD in the score of EORTC QLQ-LC13 Item 40 will be presented.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 6 years
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 4 years
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (192):
- United States (15):
  - UCLA Hematology/Oncology - Santa Monica ( Site 0023), Los Angeles, California
  - Mayo Clinic in Florida-Mayo Clinic Comprehensive Cancer Center ( Site 0001), Jacksonville, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0005), Orange City, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0003), Marietta, Georgia
  - Karmanos Cancer Institute ( Site 0018), Detroit, Michigan
  - Mayo Clinic in Rochester, Minnesota-Mayo Clinic Comprehensive Cancer Center ( Site 0027), Rochester, Minnesota
  - Hattiesburg Clinic Hematology/Oncology ( Site 0010), Hattiesburg, Mississippi
  - University Of Nebraska Medical Center ( Site 0011), Omaha, Nebraska
  - Englewood Hospital and Medical Center ( Site 0033), Englewood, New Jersey
  - Atlantic Health System Morristown Medical Center ( Site 0031), Morristown, New Jersey
  - Capital Health Medical Center - Hopewell ( Site 0006), Pennington, New Jersey
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 0015), Cincinnati, Ohio
  - Tennessee Oncology (0036), Nashville, Tennessee
  - University of Texas MD Anderson (0037), Houston, Texas
  - VCU Health Adult Outpatient Pavillion ( Site 0026), Richmond, Virginia
- Australia (4):
  - St. George Private Hospital ( Site 3004), Kogarah, New South Wales
  - Westmead Hospital ( Site 3000), Westmead, New South Wales
  - Monash Health-Oncology Research ( Site 3001), Clayton, Victoria
  - Western Health-Sunshine & Footscray Hospitals-Cancer Services-Cancer Research ( Site 3003), Melbourne, Victoria
- Brazil (6):
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0447), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0440), Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0444), Barretos, São Paulo
  - Hospital Paulistano-Americas Oncologia ( Site 0441), São Paulo
  - A. C. Camargo Cancer Center-CAPEC ( Site 0442), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0446), São Paulo
- Canada (2):
  - William Osler Health System ( Site 0205), Brampton, Ontario
  - Princess Margaret Cancer Centre ( Site 0204), Toronto, Ontario
- Chile (10):
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0501), Talca, Maule Region
  - Centro de Estudios Clínicos SAGA ( Site 0517), Santiago, Region M. de Santiago
  - Orlandi Oncologia-Oncology ( Site 0504), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0509), Santiago, Region M. de Santiago
  - K2 Oncology ( Site 0514), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 0511), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0502), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0507), Santiago, Region M. de Santiago
  - Centro Investigacion Cancer James Lind ( Site 0513), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0500), Viña del Mar, Región de Valparaíso
- China (28):
  - Anhui Provincial Cancer Hospital ( Site 2830), Hefei, Anhui
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 2810), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 2815), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital-Medical Oncology ( Site 2814), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital ( Site 2819), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 2820), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 2818), Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital-Respiratory Oncology ( Site 2816), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital-oncology of department ( Site 2807), Harbin, Heilongjiang
  - Henan Cancer Hospital-henan cancer hospital ( Site 2813), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 2805), Wuhan, Hubei
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 2806), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 2809), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University ( Site 2827), Changsha, Hunan
  - Hunan Cancer Hospital-thoracic oncology II ( Site 2808), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 2812), Nangjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Oncology Department ( Site 2821), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital-clinical research ( Site 2803), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology ( Site 2817), Xi'an, Shaanxi
  - Jinan Central Hospital-oncology department ( Site 2802), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 2804), Linyi, Shandong
  - Shanghai Chest Hospital-Oncology department ( Site 2800), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center-Oncology ( Site 2811), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University-Lung cancer center ( Site 2826), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 2822), Chengdu, Sichuan
  - Yunnan Province Cancer Hospital ( Site 2824), Kunming, Yunnan
  - Sir Run Run Shaw Hospital School of Medicine Zhejiang University ( Site 2828), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2829), Hangzhou, Zhejiang
- Czechia (5):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 1100), Brno, Brno-mesto
  - Nemocnice AGEL Ostrava - Vitkovice a.s.-Plicni odd ( Site 1103), Ostrava, Ostrava Mesto
  - Fakultni nemocnice Plzen ( Site 1104), Pilsen, Plzeň Region
  - Fakultni nemocnice Olomouc-Klinika plicnich nemoci a tuberkulozy ( Site 1102), Olomouc
  - Vseobecna fakultni nemocnice v Praze-Onkologicka klinika ( Site 1105), Prague
- France (5):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cance-Medical Oncology ( Site 1303), Bordeaux, Aquitaine
  - CENTRE LEON BERARD ( Site 1305), Lyon Cedex08, Auvergne-Rhône-Alpes
  - CHU Charles Nicolle-pneumology, intensive care and thoracic oncology ( Site 1300), Rouen, Haute-Normandie
  - Groupe hospitalier Paris saint Joseph. ( Site 1307), Paris
  - Institut Curie-Thorax Institute ( Site 1304), Paris
- Germany (6):
  - Universitaetsklinikum Freiburg ( Site 1405), Freiburg, Brandenburg
  - Universitätsmedizin Göttingen - Georg-August-Universität-Klinik für Hämatologie und Medizinische On ( Site 1407), Göttingen, Lower Saxony
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung ( Site 1400), Essen, North Rhine-Westphalia
  - Klinikum Chemnitz - Flemmingstraße ( Site 1401), Chemnitz, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden ( Site 1402), Dresden, Saxony
  - Asklepios Klinik Harburg ( Site 1403), Hamburg
- Greece (6):
  - Errikos Dunant Hospital Center-Fourth Department of Oncology and Clinical Trials Unit ( Site 2705), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 2700), Athens, Attica
  - Aretaieio Hospital ( Site 2702), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL-Oncology ( Site 2704), Chaidari, Athens, Attica
  - "Theagenio" Cancer Hospital of Thessaloniki ( Site 2703), Thessaloniki, Central Macedonia
  - Papageorgiou General Hospital of Thessaloniki ( Site 2701), Thessaloniki
- Hong Kong (4):
  - Hong Kong Integrated Oncology Centre ( Site 3200), Central
  - Queen Mary Hospital ( Site 3203), Hksar
  - Queen Elizabeth Hospital-Department of Clinical Oncology ( Site 3204), Kowloon
  - Princess Margaret Hospital-Department of Oncology ( Site 3201), Lai Chi Kok
- Israel (3):
  - Rambam Health Care Campus-Oncology Division ( Site 1702), Haifa
  - Shaare Zedek Medical Center ( Site 1700), Jerusalem
  - Rabin Medical Center ( Site 1703), Petah Tikva
- Italy (5):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 1806), Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1802), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1800), Milan, Lombardy
  - Istituto Clinico Humanitas ( Site 1803), Rozzano, Lombardy
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 2 ( Site 1805), Rome, Roma
- Japan (20):
  - Aichi Cancer Center ( Site 3400), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 3419), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 3406), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 3415), Matsuyama, Ehime
  - Gunma Prefectural Cancer Center ( Site 3418), Otashi, Gunma
  - Takarazuka City Hospital ( Site 3409), Takarazuka, Hyōgo
  - Kanazawa University Hospital ( Site 3414), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 3404), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 3416), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 3401), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 3405), Niigata, Niigata
  - Kansai Medical University Hospital ( Site 3410), Hirakata, Osaka
  - Shizuoka Cancer Center ( Site 3403), Nagaizumi-cho,Sunto-gun, Shizuoka
  - Cancer Institute Hospital of JFCR ( Site 3402), Koto, Tokyo
  - Chiba University Hospital ( Site 3411), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 3412), Fukuoka
  - Kyushu University Hospital ( Site 3407), Fukuoka
  - Okayama University Hospital ( Site 3417), Okayama
  - Osaka International Cancer Institute ( Site 3413), Osaka
  - Nippon Medical School Hospital ( Site 3408), Tokyo
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II-Medical Department ( Site 3502), Kota Bharu, Kelantan
  - National Cancer Institute-Radiotherapy and Oncology ( Site 3504), Putrajaya, Kuala Lumpur
  - Sarawak General Hospital-Radiotherapy Unit ( Site 3500), Kuching, Sarawak
- Mexico (4):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0706), Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Hematologia and Oncologia ( Site 0704), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0701), Oaxaca City, Oaxaca
  - Clinica Integral Internacional de Oncología ( Site 0705), Puebla City
- Philippines (6):
  - THE MEDICAL CITY ILOILO-The Medical City Iloilo - Clinical and Translational Research Institute-Ilo ( Site 3600), Iloilo City, Iloilo
  - Manila Doctors Hospital-Clinical Trial Office ( Site 3604), Manila, National Capital Region
  - Asian Hospital and Medical Center ( Site 3605), Muntinlupa, National Capital Region
  - THE MEDICAL CITY-Cancer Research Center ( Site 3603), Pasig, National Capital Region
  - ST. LUKE'S MEDICAL CENTER ( Site 3601), Quezon City, National Capital Region
  - CARDINAL SANTOS MEDICAL CENTER-Research Room ( Site 3602), San Juan City, Metro Manila, National Capital Region
- Poland (7):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2003), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Zespolony im Ludwika Rydygiera w Toruniu ( Site 2009), Torun, Kuyavian-Pomeranian Voivodeship
  - Instytut Gruźlicy i Chorób Płuc w Warszawie ( Site 2011), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2000), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 2001), Przemyśl, Podkarpackie Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-II Klinika Radioterapi i Chemioterapii ( Site 2002), Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 2005), Kielce, Świętokrzyskie Voivodeship
- South Korea (14):
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 3807), Hwasun, Jeonranamdo
  - National Cancer Center-Lung Cancer Center ( Site 3810), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 3806), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 3803), Suwon, Kyonggi-do
  - Pusan National University Yangsan Hospital-Lung Cancer Clinic ( Site 3811), Yangsan, Kyongsangnam-do
  - Chungbuk National University Hospital-Internal medicine ( Site 3809), Cheongju-si, North Chungcheong
  - Pusan National University Hospital ( Site 3805), Busan, Pusan-Kwangyokshi
  - Chungnam national university hospital ( Site 3808), Junggu, Taejon-Kwangyokshi
  - Kangbuk Samsung Hospital ( Site 3813), Seoul
  - Severance Hospital, Yonsei University Health System-Lung Cancer Center ( Site 3804), Seoul
  - Konkuk University Medical Center ( Site 3812), Seoul
  - Asan Medical Center ( Site 3801), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3802), Seoul
  - Korea University Guro Hospital-Internal Medicine ( Site 3800), Seoul
- Spain (7):
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 2304), Barcelona, Catalonia
  - Hospital Insular de Gran Canaria-Oncology ( Site 2305), Las Palmas de Gran Canaria, Las Palmas
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2301), Pozuelo de Alarcón, Madrid
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 2303), Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General-Oncology ( Site 2302), Málaga, Malaga
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2300), Barcelona
  - Clinica Universidad de Navarra-Medical Oncology ( Site 2306), Madrid
- Taiwan (11):
  - Chi Mei Medical Center ( Site 3910), Tainan, Tainan
  - National Taiwan University Cancer Center (NTUCC) ( Site 3903), Taipei City, Taipei
  - Changhua Christian Hospital ( Site 3908), Changhua
  - National Taiwan University Hospital - Hsinchu branch ( Site 3907), Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 3912), Kaohsiung City
  - E-Da hospital ( Site 3911), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3906), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 3909), Tainan
  - National Taiwan University Hospital-Oncology ( Site 3904), Taipei
  - Mackay Memorial Hospital-Chest Medicine ( Site 3902), Taipei
  - Taipei Medical University Hospital ( Site 3900), Taipei
- Thailand (6):
  - Faculty of Medicine Siriraj Hospital ( Site 4000), Bangkok, Bangkok
  - Lampang Cancer Hospital ( Site 4005), Muang, Changwat Lampang
  - Songklanagarind hospital ( Site 4001), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 4003), Muang, Chiang Mai
  - Faculty of Medicine - Khon Kaen University ( Site 4004), Khon Kaen
  - Sunpasitthiprasong Hospital-Oncology ( Site 4002), Ubon Ratchathani
- Turkey (Türkiye) (6):
  - Medipol Mega Universite Hastanesi-oncology ( Site 2505), Stanbul, Istanbul
  - Ege Universitesi Hastanesi-Chest Diseases Department ( Site 2504), Bornova, İzmir
  - Adana Medical Park Seyhan Hastanesi ( Site 2506), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2500), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 2501), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2502), Istanbul
- United Kingdom (6):
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 2606), London, Kensington and Chelsea
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 2600), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust-Oncology & Haematology Clinical Trials ( Site 2603), London, London, City of
  - Royal Marsden Hospital (Sutton) ( Site 2605), Sutton, Surrey
  - The Christie NHS Foundation Trust ( Site 2604), Manchester
  - The Clatterbridge Cancer Centre ( Site 2602), Metropolitan Borough of Wirral
- Vietnam (3):
  - Hanoi Oncology Hospital ( Site 4102), Hanoi, Hanoi
  - K Hospital - National Cancer Hospital ( Site 4105), Hanoi, Hanoi
  - National Lung Hospital-Oncology Department ( Site 4104), Hanoi, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26168&tenant=MT_MSD_9011